CLINICAL TRIAL: NCT03961659
Title: A Prospective, Randomized, Open Label, Parallel, 16-week Study to Explore and Evaluate the Therapeutic Effects of Liraglutid, Dapagliflozin and Acarbose on the Cognitive Function, Olfactory Function, and Odor-induced Brain Activation in Overweight/Obese Patients With T2DM Inadequately Controlled With Metformin Monotherapy.
Brief Title: Effects of Liraglutid, Dapagliflozin and Acarbose on the Cognitive Function, Olfactory Function, and Odor-induced Brain Activation in Overweight/Obese T2DM Patients Controlled Inadequately With Metformin Monotherapy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Dalong Zhu, Chief Physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZZ2019
Record Dates: First submitted 2019-05-19; First posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Type 2 Diabetes Mellitus; Obesity; Cognitive Impairment
Keywords: Functional MRI; Olfactory function; Liraglutid; Dapagliflozin; Acarbose
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Cognitive Dysfunction | interventions — Metformin; dapagliflozin; Acarbose

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Liraglutid (Active Comparator): Liraglutid will be titrated from 0.6mg/day to a final dose 1.8mg/day during the first 2 weeks, if well tolerated. Meanwhile, All patients will also continue on their existing dose and regimen of metformin throughout the study. Visits at 4-week intervals will be performed to evaluate the safety of drugs. Metformin dose can be reduced in response to hypoglycaemia, but liraglutid could not be adjusted. If the plasma glucose still not achieve the target at the maximum dose, the maximum dose will be maintained until the completion of the study.
  Interventions: Drug: Liraglutid
- Dapagliflozin (Active Comparator): Dapagliflozin will be initiated and maintained at 10mg/day every morning until the completion of the study. Meanwhile, All patients will also continue on their existing dose and regimen of metformin throughout the study. Visits at 4-week intervals will be performed to evaluate the safety of drugs. Metformin dose can be reduced in response to hypoglycaemia, but dapagliflozin could not be adjusted. If the plasma glucose still not achieve the target at the maximum dose, the maximum dose will be maintained until the completion of the study.
  Interventions: Drug: Dapagliflozin
- Acarbose (Active Comparator): Acarbose will be initiated at 50mg three times daily for the first week, and then titrated to100mg three times daily if appropriate. Meanwhile, All patients will also continue on their existing dose and regimen of metformin throughout the study. Visits at 4-week intervals will be performed to evaluate the safety of drugs. Metformin dose can be reduced in response to hypoglycaemia, but acarbose could not be adjusted. If the plasma glucose still not achieve the target at the maximum dose, the maximum dose will be maintained until the completion of the study.
  Interventions: Drug: Acarbose

INTERVENTIONS:
Drug: Liraglutid — Liraglutid will be titrated from 0.6mg/day to 1.8mg/day during the first 2 weeks, if well tolerated. All patients will also continue on their existing dose and regimen of metformin throughout the study.
  Other Names: metformin
  Arms: Liraglutid
Drug: Dapagliflozin — Dapagliflozin will be initiated and maintained at 10mg/day every morning until the completion of the study. All patients will also continue on their existing dose and regimen of metformin throughout the study.
  Other Names: metformin
  Arms: Dapagliflozin
Drug: Acarbose — Acarbose will be initiated at 50mg three times daily for the first week, and then titrated to 100mg three times daily if appropriate.All patients will also continue on their existing dose and regimen of metformin throughout the study.
  Other Names: metformin
  Arms: Acarbose

SUMMARY:
This is a prospective, randomized, open label, parallel, 16-week study to explore and evaluate the therapeutic effects of liraglutid, dapagliflozin and acarbose on the cognitive function, olfactory function, and odor-induced brain activation in overweight/obese patients with type 2 diabetes mellitus(T2DM) inadequately controlled with metformin monotherapy.

DETAILED DESCRIPTION:
This is a prospective, randomized, open label, parallel, 16-week study to explore and evaluate the therapeutic effects of liraglutid, dapagliflozin and acarbose on the cognitive function, olfactory function, and odor-induced brain activation in overweight/obese patients with T2DM inadequately controlled with metformin monotherapy.We have 1 principle investigator, 6 sub-investigators and 1 nurse in research centre. The sub-investigators will screen in the outpatient and inpatient departments to enroll 87 patients (29 for each arm) totally with the inclusion and exclusion criteria in 12 months. The patients will be randomized at a 1:1:1 ratio into liraglutid, dapagliflozin and acarbose treatment group with a computer-generated random order. All patients will also continue on their existing dose and regimen of metformin throughout the study. At the baseline, clinical information collection, 100g-steamed bread meal test, biochemical measurement, body composition analysis, cognitive assessment, olfactory test and functional magnetic resonance imaging(fMRI) scan will be conducted for all patients. During the treatment period, visits at 4-week intervals will be performed to evaluate the safety of drugs and adjust the dose of metformin if hypoglycaemia occurs; meanwhile, fasting and 2-hour postprandial plasma glucose assayed by fingerstick, physical examination, and olfactory test will be conducted. At the end of the study, all of the assessments will be performed again for all recruited subjects, including early withdrawal patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≧ 40 and ≦75 years old
* T2DM patients controlled with metformin monotherapy with stable, maximum tolerated doses (≧1500mg/d, ≧12 weeks)
* HbA1c>7% and ≤9%
* Body mass index(BMI) ≥25kg/m2 and with stable weight during previous 3 months
* Right handedness
* Possessed over 6-year education
* Provision of informed consent prior to any study specific procedures
* Mini-Mental State Examination (MMSE) >24

Exclusion Criteria:

* Allergies to research drugs
* Treated with glucagon-like peptide-1 receptor agonists, dipeptidyl peptidase-4 inhibitors, sodium-glucose cotransporter 2 inhibitors, insulins, and glycosidase inhibitors in the previous 6 months
* Moderate to severe renal dysfunction defined as estimated glomerular filtration rate(eGFR)<60ml/min/1.73m2 ( eGFR was estimated by CKD-EPI creatinine equation using an online calculator).
* Hepatic insufficiency
* A history of neurological and psychiatric disorders, nasal pathologies, abnormal thyroid, pancreatitis, repeated urinary tract infection, chronic gastrointestinal dysfunction, any disease that may worsen by intestinal flatulence, alcohol or substance abuse, steroid treatment
* Any acute disease
* Inability to undergo tests or MRI scanning
* Pregnant or lactating women
* Participating in other clinical trials at the same time or within 6 months prior to the start of the trial

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Change of olfactory brain activation by fMRI | from baseline to 16 weeks' follow-up.
  Compare the change of olfactory brain activation by fMRI from baseline to 16 weeks' follow-up

SECONDARY OUTCOMES:
Change of cognitive function | from baseline to 16 weeks' follow-up.
  Compare the change of Montreal Cognitive Assessment (MoCA, beijing version) from baseline to 16 weeks' follow-up. MoCA score(ranging from 0 to 30)<26 is considered cognitive impairment and when the score is lower, the cognitive impairment is more serious. MoCA score ≥26 is considered normal cognition.
Proportion of patients whose MoCA<26 scores | at baseline and at 16 weeks' follow-up.
  Compare the proportion of patients whose MoCA<26 scores at baseline and at 16 weeks' follow-up.
Change of blood glycaemic control | from baseline to 16 weeks' follow-up
  Compare the change of glycosylated hemoglobin(HbA1c) from baseline to 16 weeks' follow-up
Proportion of patients whose HbA1c<7% | at 16 weeks' follow-up.
  Analyze the proportion of patients whose HbA1c<7% at 16 weeks' follow-up.
Proportion of patients whose weight loss>3% and >5% | from baseline to 16 weeks' follow-up.
  Analyze the proportion of patients whose weight loss>3% and >5%
Olfactory threshold test | from baseline to 16 weeks' follow-up.
  The olfactory threshold test (score range 1-13.5) is determined based on a series of binary dilutions of the N-butanol solution in light mineral oil. The higher the score is, the more sensitive the participant is in detecting an odor. Scores of 8-10 were considered normal olfactory sensitivity, whereas scores of 1-3 signified olfactory dysfunction or anosmia, and scores of ≥10 indicate better olfactory sensitivity.

CONTACTS AND LOCATIONS:
Locations (1):
- at Division of Endocrinology, the Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Cheng H, Zhang Z, Zhang B, Zhang W, Wang J, Ni W, Miao Y, Liu J, Bi Y. Enhancement of Impaired Olfactory Neural Activation and Cognitive Capacity by Liraglutide, but Not Dapagliflozin or Acarbose, in Patients With Type 2 Diabetes: A 16-Week Randomized Parallel Comparative Study. Diabetes Care. 2022 May 1;45(5):1201-1210. doi: 10.2337/dc21-2064. PMID 35263425